CLINICAL TRIAL: NCT01522755
Title: Predictive Factors of a Successful Implant of the CapsureFix MRI Model 5086
Status: Completed | Type: Observational
Sponsor: Medtronic Cardiac Rhythm and Heart Failure (Industry)
Collaborators: Medtronic (Industry)
Responsible Party: Sponsor
Other Study IDs: 11
Record Dates: First submitted 2012-01-11; First posted 2012-02-01 (Estimated); Results first posted 2020-01-18 (Actual); Last update posted 2025-07-02 (Actual); Status verified 2020-01

CONDITIONS: Bradyarrhythmia
Keywords: Pacing lead; implant; pacemaker
MeSH Terms: conditions — Bradycardia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients implanted with the CapsureFix MRI pacing lead: Patients implanted with the CapsureFix MRI pacing lead model 5086
  Interventions: Device: Pacing system implant with the CapsureFix MRI pacing lead model 5086

INTERVENTIONS:
Device: Pacing system implant with the CapsureFix MRI pacing lead model 5086 — Pacing system implant with the CapsureFix MRI pacing lead model 5086

SUMMARY:
Pacing leads are key elements of a pacing system as their proper functioning is one of the major factors affecting the long term performance of the whole system.

Success of a pacing lead implant can be defined considering 3 items: ease of lead implant, lead stability and lead electrical performances.

These factors may be related to the physician experience (global implant experience, experience with a given lead), to the implant procedure (lead access, lead position, implant time, scopy time) to the lead (handling and mechanical characteristics) and to the patient (ischemic history).

Even though implant success rate is quite high with currently available leads, the weight of the different factors influencing success has never been studied systematically. The objective of the current study is then to define the predictive factors of an implant success with the CapsureFix MRI model 5086.

This lead has been selected because it has been available for a short period, so the investigators have a limited experience of it and it has a unique design which makes it conditionally safe in an MRI environment and which may be associated with specific handling characteristics.

ELIGIBILITY:
Inclusion Criteria:

* Patient older than 18
* Patient implanted with a fully automatic ICD and remotely followed-up,
* Patient geographically stable and able to attend FU at investigative site
* Patient who signed a data release authorization form,

Exclusion Criteria:

* Patient whose mental or physical capacity impedes to give an informed data release authorization,
* Patient already enrolled in a clinical study whose procedures may interfere with the results of the present study,
* Patients in New York Heart Association (NYHA) class IV

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient implanted with 2 CapsureFix MRI pacing leads model 5086 in the atrium and in the ventricle
Sampling Method: Non-Probability Sample
Enrollment: 409 (Actual)
Dates: Start 2011-05; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Olivier BIZEAU, MD, Principal Investigator — Centre Hospitalier Regionnal d'Orléans La Source
Locations (1):
- Centre Hospitalier Regionnal d'Orléans La Source, Orléans, France

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment period: 31 January 2010 - 24 January 2013. 32 implanting centers and 41 implanters participated in the study.
Period: Overall Study
Arm/Group | Patients Implanted With the CapsureFix MRI Pacing Lead
Started | 409
Completed | 409
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Patients Implanted With the CapsureFix MRI Pacing Lead
Number analyzed (Participants) | 409
Age, Continuous [Mean (Standard Deviation); unit: years] | 72.5 (10.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 151
  Male | 258
Region of Enrollment [Number; unit: participants]
  France | 409
Pacing indication [Number; unit: participants]
  Sinoatrial block | 40
  Sinus bradycardia | 51
  1st degree AV block | 21
  2nd degree AV block Wenckebach | 19
  2nd degree AV block Mobitz 2 | 62
  Permanent 3rd degree AV block | 59
  Paroxysmal 3rd degree AV block | 57
  Sinus node disease | 82
  Other | 18
Atrial arrhythmia history [Number; unit: participants]
  Patients with atrial arrhythmia history | 126
  Patients with no atrial arrythmia history | 283
Ventricular arrhythmia history [Number; unit: participants]
  Patients with ventricular arrhytmia history | 14
  Patients with no ventricular arrhythmia history | 395
cardiac disease history [Number; unit: participants]
  Patients with cardiac disease history | 95
  Patient with no cardiac disease history | 314
coronary disease history [Number; unit: participants]
  Patients with coronary disease history | 59
  Patients with no coronary disease history | 350
Myocardial infarction history [Number; unit: participants]
  Patients with myocardial infarction history | 28
  Patients with no myocardial infarction history | 381
Stroke history [Number; unit: participants]
  Patients with stroke history | 37
  Patients with no stroke history | 372

OUTCOME MEASURES:

1. Primary Outcome: Ease of Implant
Description: Ease of implant as experienced by the implanting physician on maneuverability of the catheter. This was measured by a questionnaire for which each criterion was coded as Very Good, Good, Fair, Poor, Very Poor. Coding 9, 7, 5, 3, 1 was applied for each response with 9 representing Very Good. An average was calculated for each evaluation and for each probe implantation site.
Time Frame: at implant
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Implanting Physicians: Questionnaires on ease of implant, maneuverability of the catheter, and other variables were taken during this study.
Arm/Group | Implanting Physicians
Number analyzed (Participants) | 41
score on a scale
  maneuverability for the atrium | 6.9 (1.2)
  maneuverability for the ventricle | 6.3 (1.0)

2. Primary Outcome: Lead Stability
Description: Lead stability of the Capsure Fix as measured by number of dislodgments
Time Frame: 3 months
Measure: Number; unit: dislodgements
Arm/Group | Patients Implanted With the CapsureFix MRI Pacing Lead
Number analyzed (Participants) | 409
dislodgements | 10

3. Primary Outcome: Pacing Threshold During and Post Implant of the CapsureFix MRI Lead Model 5086
Description: Change of pacing threshold will be measured during and post implant of the CapsureFix MRI lead model 5086
Time Frame: 3 months
Population: 409 patients have been consecutively enrolled in 32 sites.
Measure: Mean (Standard Deviation); unit: Volt
Arm/Group | Patients Implanted With the CapsureFix MRI Pacing Lead
Number analyzed (Participants) | 409
Volt
  Pacing threshold Implant (RA) | 0.9 (0.5)
  Pacing threshold Post implant (RA) | 0.6 (0.3)
  Pacing threshold Implant (RV) | 0.7 (0.4)
  Pacing threshold Post implant (RV) | 0.6 (0.3)
Statistical Analysis 1: Comparison: Patients Implanted With the CapsureFix MRI Pacing Lead; Test type: Other — t-test; p < 0.05, t-test, 2 sided

4. Primary Outcome: Sensing Amplitude During and Post Implant of the CapsureFix MRI Lead Model 5086
Description: Change of sensing amplitude will be measured during and post implant of the CapsureFix MRI Lead Model 5086
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: mV
Arm/Group | Patients Implanted With the CapsureFix MRI Pacing Lead
Number analyzed (Participants) | 409
mV
  Sensing Implant (RA) | 3.2 (1.9)
  Sensing Post Implant (RA) | 3.2 (2.2)
  Sensing Implant (RV) | 10.9 (5.2)
  Sensing Post Implant (RV) | 9.5 (4.5)
Statistical Analysis 1: Comparison: Patients Implanted With the CapsureFix MRI Pacing Lead; Test type: Other — t-test; p < 0.05, t-test, 2 sided

5. Primary Outcome: Impedance Measurements During and Post Implant of the CapsureFix MRI Lead Model 5086
Description: Change of impedance will be measured during and post implant of the CapsureFix MRI Lead Model 5086
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: Ohm
Arm/Group | Patients Implanted With the CapsureFix MRI Pacing Lead
Number analyzed (Participants) | 409
Ohm
  Impedance Implant RA | 704 (242)
  Impedance Post Implant RA | 547 (175)
  Impedance Implant RV | 896 (286)
  Impendance Post Implant RV | 635 (200)
Statistical Analysis 1: Comparison: Patients Implanted With the CapsureFix MRI Pacing Lead; Test type: Other — t-test; p < 0.05, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: From the informed consent signature to the end of the study.
Arm/Group | Patients Implanted With the CapsureFix MRI Pacing Lead
Serious Adverse Events (participants affected / at risk) | 16/409
Other Adverse Events (participants affected / at risk) | 11/409
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Patients Implanted With the CapsureFix MRI Pacing Lead (N=409)
Lead displacement (Cardiac disorders) | 10 (10)
hemopericardium (Cardiac disorders) | 2 (2)
Hospitalization (Cardiac disorders) | 1 (1)
Permanent disability (Musculoskeletal and connective tissue disorders) | 1 (1)
Hospitalization due to electrical issue (Cardiac disorders) | 2 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Patients Implanted With the CapsureFix MRI Pacing Lead (N=409)
electrical abnormal parameters (Cardiac disorders) | 8 (8)
lead displacement (Cardiac disorders) | 2 (2)
pneumothorax (Cardiac disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No